CLINICAL TRIAL: NCT00636363
Title: Safety and Efficacy of a Bausch & Lomb Multipurpose Solution When Compared to Ciba Vision Aquify Multipurpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 554
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Contact Lens Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multipurpose Solution - Rub Care (Experimental): Bausch & Lomb Multipurpose Solution for use with contact lens care
  Interventions: Device: Bausch & Lomb Multipurpose Solution - Rub Care
- Multipurpose Solution - No Rub Care (Experimental): Bausch & Lomb Multipurpose Solution for use with contact lens care
  Interventions: Device: Bausch & Lomb Multipurpose Solution - No Rub Care
- Ciba Vision Aquify Multipurpose Solution (Active Comparator): Ciba Vision Aquify Multipurpose Solution for use with contact lens care
  Interventions: Device: Ciba Vision Aquify Multipurpose Solution

INTERVENTIONS:
Device: Bausch & Lomb Multipurpose Solution - Rub Care — Daily care for contact lenses - rub care regimen
  Arms: Multipurpose Solution - Rub Care
Device: Bausch & Lomb Multipurpose Solution - No Rub Care — Daily care for contact lenses - no rub care regimen
  Arms: Multipurpose Solution - No Rub Care
Device: Ciba Vision Aquify Multipurpose Solution — daily care for contact lenses
  Arms: Ciba Vision Aquify Multipurpose Solution

SUMMARY:
To the safety and efficacy of a Bausch & Lomb Multipurpose Solution when compared to Ciba vision Aquify Multipurpose solution

ELIGIBILITY:
Inclusion Criteria:

* subject is a habitual wearer of a silicone hydrogel or group IV contact lens
* VA correctable to 0.3 LogMar or better (driving vision)
* Clear central cornea
* Subject uses a lens care system on a regular basis

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using systemic or topical medications
* wear monovision, multifocal or toric contact lenses
* Any grade 2 or greater slit lamp findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohinder Merchea, OD, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Place Eye Care, Le Roy, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 541 participants were enrolled in this 3 month study (1152 eyes). First participant was enrolled Mar 7, 2008 and last participant exited Aug 1, 2008. Participant were enrolled from 24 investigative sites in the US.
Pre-assignment Details: Of the 541 participants enrolled 6 were ineligible at baseline. These subjects met the exclusion criteria. 535 participants participated in the study.
Period: Overall Study
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution
Started | 178 | 176 | 181
Completed | 165 | 156 | 163
Not Completed | 13 | 20 | 18
Not completed — Conjunctivitis | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Positive slit lamp finding | 0 | 2 | 1
Not completed — Study related symptoms/complaints | 8 | 7 | 4
Not completed — Met ineligibility criteria | 0 | 0 | 3
Not completed — Missed > 1 visit | 0 | 1 | 3
Not completed — Lack of motivation | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Lost to Follow-up | 3 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution | Total
Number analyzed (Participants) | 178 | 176 | 181 | 535
Age, Customized [Number; unit: Participants]
  18-66 years of age | 178 | 176 | 181 | 535
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 133 | 126 | 383
  Male | 54 | 43 | 55 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 7 | 21
  Not Hispanic or Latino | 168 | 172 | 174 | 514
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 178 | 176 | 181 | 535

OUTCOME MEASURES:

1. Primary Outcome: Slit-lamp Findings > Grade 2
Description: eyes with any slit lamp findings greater than Grade 2 at any visit. Slit lamp findings for each eye will be graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). Epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, superior tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates will be assessed.
Time Frame: Over 4 visits for 3 month period
Population: Over all follow-up visits, all dispensed eyes
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution
Number analyzed (Participants) | 177 | 176 | 179
Number analyzed (eyes) | 354 | 352 | 358
participants | 3 | 4 | 3

2. Primary Outcome: Subjective Responses to Comfort Related Symptoms/Complaints
Description: Subject symptoms/complaints will be assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints.
Time Frame: Over 4 visits for the 3 month period
Population: Comfort related symptoms/complaints for all eligible, dispensed eyes. Over all follow-up visits.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Units Other Than Participants: eyes
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution
Number analyzed (Participants) | 176 | 172 | 176
Number analyzed (eyes) | 352 | 344 | 352
Scores on a Scale
  Comfort | 88.7 (12.9) | 84.6 (16.5) | 86.9 (13.9)
  End of day comfort | 83.2 (17.6) | 77.1 (20.8) | 79.1 (18.6)
  Burning/stinging upon inserstion | 91.1 (13.5) | 89.1 (15.8) | 90.1 (15.9)
  Irritation | 88.7 (15.3) | 85.0 (17.4) | 86.8 (15.2)
  Itching | 91.6 (12.7) | 90.9 (12.9) | 90.8 (14.1)
  Dryness | 88.2 (14.0) | 83.0 (19.0) | 83.7 (16.4)
  Redness | 91.4 (13.2) | 91.0 (13.1) | 91.2 (14.0)
  Vision | 91.9 (10.9) | 88.9 (16.2) | 92.6 (10.9)
  Lens cleanliness | 92.2 (11.7) | 89.2 (15.3) | 91.8 (10.8)
  Lens Handling | 95.1 (9.0) | 95.1 (7.2) | 94.9 (8.5)

3. Primary Outcome: Contact Lens Deposits
Description: Lens deposits assessed at each follow-up visit. Degree of deposits assessed as none, light, medium, or heavy.
Time Frame: At each visit for 3 months
Population: Lens deposits, All eligible, dispensed eyes.
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution
Number analyzed (Participants) | 175 | 169 | 175
Number analyzed (eyes) | 350 | 338 | 350
Eyes
  None | 98 | 52 | 91
  Light | 147 | 176 | 178
  Medium | 84 | 84 | 69
  Heavy | 21 | 26 | 12

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Multipurpose Solution - Rub Care | Multipurpose Solution - No Rub Care | Ciba Vision Aquify Multipurpose Solution
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/176 | 0/181
Other Adverse Events (participants affected / at risk) | 0/178 | 0/176 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.